CLINICAL TRIAL: NCT05000671
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Continuous Intravenous Infusion of STC314 Injection in Chinese Patients With Acute Respiratory Distress Syndrome
Brief Title: A Study to Evaluate the Safety and Effect of STC314 Injection Continuous Infusion in Subjects With Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grand Medical Pty Ltd. (Industry)
Collaborators: Grand Pharmaceutical (China) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GPHIP-0103
Record Dates: First submitted 2021-07-27; First posted 2021-08-11 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — STC3141

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Drug: STC314/Placebo injection Continuous infusion at rate 58.3mg/hr up to 3 days (72 hours) N=8(Randomization-STC314/Placebo injection=3:1)
  Interventions: Drug: STC314 injection or Placebo(rate=58.3 mg/hr)
- Cohort 2 (Experimental): Drug: STC314/Placebo injection Continuous infusion at rate 87.5mg/hr up to 3 days (72 hours) N=8(Randomization-STC314/Placebo injection=3:1)
  Interventions: Drug: STC314 injection or Placebo(rate=87.5 mg/hr)

INTERVENTIONS:
Drug: STC314 injection or Placebo(rate=58.3 mg/hr) — To receive continuous infusion of STC314/Placebo injection at rate 58.3mg/hr up to 3 days (72hours). Also to receive appropriate standard of care.
  Arms: Cohort 1
Drug: STC314 injection or Placebo(rate=87.5 mg/hr) — To receive continuous infusion of STC314/Placebo injection at rate 87.5mg/hr up to 3 days (72hours). Also to receive appropriate standard of care.
  Arms: Cohort 2

SUMMARY:
This study is a Randomized, Double-blinded, Placebo-controlled Phase Ib Study to Evaluate the Safety, Tolerability and Pharmacokinetics of STC314 Injection Administered as Continuous Intravenous Infusion in Chinese Patients with ARDS (Acute Respiratory Distress Syndrome).

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 70 years, male or female;
2. Voluntarily participate in the study and sign the informed consent form;
3. Diagnosis of ARDS for no more than 48 hours (starting at the time of diagnosis recorded in the medical record)；
4. The following 2012 Berlin definition criteria for mild to moderate ARDS were met:

   1. From known clinical impairment and new or worsening of respiratory symptoms to fulfillment of diagnostic criteria is less than 7 days(inclusive).
   2. Chest imaging suggests bilateral infiltrates. The effusion, lobar/atelectasis, or nodules cannot completely explain the phenomenon.
   3. Respiratory failure cannot be completely explained by heart failure or fluid overload;
   4. When PEEP or CPAP ≥5 cm H2O, 100 mmHg≤PaO2/FiO2≤300 mmHg;
5. Male subjects agree to use an effective contraceptive method from the start of the study until 7 days after the end of treatment; Female subjects of childbearing age agree to use an effective contraceptive method from the start of the study until 3 months after the end of treatment.

Exclusion Criteria:

1. Positive serum pregnancy test before dosing for women of childbearing potential, pregnant women, or lactating women;
2. Terminal phase of chronic disease with an expected survival of no more than 6 months;
3. Combined with one of the following chronic organ damage or immunosuppressive diseases:

   1. Heart: New York Heart Association functional class IV;
   2. Lung: severe lung disease, including pulmonary hypertension, oxygen therapy or ventilator dependence for more than one month cumulatively within the first six months of screening, end-stage lung disease, or severe exercise limitation caused by chest wall malformations;
   3. Kidney: ongoing long-term dialysis treatment;
   4. Liver: biopsy confirmed cirrhosis and portal hypertension, or previous upper gastrointestinal bleeding caused by portal hypertension; Liver failure, hepatic encephalopathy, or hepatic coma;
   5. Immunosuppression: with lymphoma, leukemia or acquired immunodeficiency; Received anti-tumor chemotherapy in the last 3 months, or ongoing immunosuppressive therapy due to organ transplantation, immune diseases, etc.; Has undergone allogeneic bone marrow transplantation or hematopoietic stem cell transplantation; Steroid hormone therapy in the last 3 months (equivalent to > 0.5 mg/kg/day prednisone continued 1 month);
4. History of one of the following within 4 weeks prior to screening:

   1. Acute pulmonary embolism;
   2. Cardiac arrest;
   3. Acute myocardial infarction;
5. eGFR < 60 mL/min/BSA (calculated using CG formula);
6. ALT > 5 x ULN, or total bilirubin > 2 x ULN;
7. Severe anemia (hemoglobin < 7.0 g/dL);
8. Absolute neutrophil count < 1500/μL;
9. Platelet count < 50,000/μL;
10. aPTT > 1.5 × ULN;
11. Active bleeding that cannot be effectively controlled;
12. The subject required therapeutic doses of heparin or was taking anticoagulants;
13. ARDS caused by direct lung injury due to physical or chemical causes;
14. Severe or greater burns: the overall surface area of burns exceeds 30% or the III degree burn area exceeds 10%; or the total area is less than 30%, but the general condition is severe or has shock, combined injury, respiratory tract burn;
15. Allergic to the active ingredients or excipients of the study drug;
16. Subjects have participated in other clinical studies (other than those who have not received intervention) or are participating in other experimental treatments within 1 month prior to screening;
17. In the opinion of the investigator, the subject could not benefit from the study or was not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  The incidence of adverse event (AE) and serious adverse event (SAE);
To evaluate the safety of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Rates of Treatment Discontinuation Due to Adverse Events;
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  maximum concentration (Cmax)
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  area under the plasma concentration-time curve (AUC0-t, AUC0-inf)
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  time to peak (Tmax)
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  elimination half Decay (t1/2)
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  elimination rate constant(Kel)
To evaluate the pharmacokinetic of STC314 injection in patients with ARDS. | Through 0 to144 hours after the start of treatment
  clearance (CL)

SECONDARY OUTCOMES:
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Changes of the value of blood lactate from baseline after dosing
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of Oxygenation Index (PaO2/FiO2) from baseline after dosing
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of Murray Lung Injury Score from baseline.(range 0-4, higher score means more severe lung injury)
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of the value of serum creatinine from baseline after dosing
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of the value of bilirubin from baseline after dosing
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of the value of Alanine Transaminase(ALT) from baseline after dosing
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Change of Sequential Organ Failure Assessment score from baseline after dosing.(range 0-4, higher score means a worse prognosis)
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  all-cause mortality within 28 days
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Ventilator-free survival time within 28 days
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  Hospitalization time within 28 days
To evaluate the efficacy of STC314 injection in patients with ARDS. | Within 28 days after the start of treatment
  length of ICU stay within 28 days

OTHER OUTCOMES:
As an exploratory objective, the change in biomarkers from baseline following STC314 injection treatment in subjects with Acute Respiratory Distress Syndrome will be evaluated. | Through 0 to144 hours after the start of treatment
  Change of the level of Histone in plasma after dosing
As an exploratory objective, the change in biomarkers from baseline following STC314 injection treatment in subjects with Acute Respiratory Distress Syndrome will be evaluated. | Through 0 to144 hours after the start of treatment
  Change of the level of Neutrophil extracellular traps(NETs)-related variables in plasma after dosing [myelinated Oxidase (MPO), citrullinated histone H3 (CitH3), circular free DNA (cfDNA)]
As an exploratory objective, the change in biomarkers from baseline following STC314 injection treatment in subjects with Acute Respiratory Distress Syndrome will be evaluated. | Through 0 to144 hours after the start of treatment
  Change of the level of inflammatory factor interleukin-6 (IL-6) after dosing

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Jinyintan Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No